CLINICAL TRIAL: NCT04422483
Title: A Realist Evaluation of Autism ServiCe Delivery (RE-ASCeD): Which Diagnostic Pathways Work Best, for Whom, When, and at What Cost?
Brief Title: A Realist Evaluation of Autism ServiCe Delivery (RE-ASCeD)
Acronym: Re-ASCed
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sussex Community NHS Foundation Trust (Other)
Collaborators: University of Kent (Other); University of Surrey (Other); Newcastle University (Other); Council for Disabled Children (Unknown); Autistica (Unknown); West Sussex Parent Carer Forum (Unknown); Northumberland, Tyne and Wear NHS Foundation Trust (Other); Cambridgeshire and Peterborough NHS Foundation Trust (Other); Brighton & Sussex Medical School (Other); National Health Service, United Kingdom (Other Government)
Responsible Party: Principal Investigator, William Farr, Principal Investigator, Sussex Community NHS Foundation Trust
Other Study IDs: Re-ASCed Protocol IM 17-4-20
Record Dates: First submitted 2020-05-18; First posted 2020-06-09 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Autism; Children; Family; Diagnoses, Syndromes, and Conditions; Patient Satisfaction
MeSH Terms: conditions — Autistic Disorder; Disease; Patient Satisfaction | interventions — Focus Groups; Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Service Model Level Case Studies: Realist Interviews. MONTHS 9-30 (N=6-8 sites, 12 people per site, 96 interviewees)
  Interventions: Other: Realist evaluation
- Individual/family level interviews: Child Interviews. MONTHS 9-30 (N=6-8 sites, 6 people per site, max. 48 interviewees)
  Interventions: Other: Realist evaluation
- Individual child/family Level Case Studies:: MONTHS 10-30 (N=6-8 sites, 78 people per model (x4), 312 participants, 156 per NU/SCFT depending on distribution of sites)
  Interventions: Other: Realist evaluation
- Focus groups:: MONTHS 9-30 (N=6-8 sites, 6-8 focus groups of up to 8 parents) N= 64
  Interventions: Other: Realist evaluation

INTERVENTIONS:
Other: Realist evaluation — In-depth exploration of individual service models will be carried out to determine the interrelationship of context, intervention, mechanisms and outcomes as they occur in their natural setting. Data will be gathered within case studies using mixed methods at two levels: (i) service model and (ii) individual child/ family. Methods will include semi structured realist Interviews, focus groups, and document reviews to assemble a comprehensive description of the service and model. Interviewees will include commissioners, service managers, clinicians, referrers, parents and young people. Interviews will be recorded and transcribed, proceeding to qualitative analysis based on components of the programme theory. Regular team meetings will discuss coding, address inconsistencies, and refine collective understanding of coding framework. Coded data will be collated using NVivo software.
  Other Names: focus group; health economic questionnaire; survey; Interview; Case note data

SUMMARY:
Diagnostic pathways for children with possible autism. Which work best, for whom, when, and at what cost? Autism is a complex neuro-behaviour condition. People with autism have difficulty with social interaction and in communication with others. They may struggle with change, and repeat actions over and over. Life may be very anxious or stressful. The signs of autism can occur at any age but often appear in the first two years of life. There is no one type of autism, but many, so the condition is now called autism spectrum disorder (ASD). Autism is lifelong but this study is only about children. Caring for a child with autism can be difficult and can sometimes be tough on the whole family.

This project aims to guide the people who plan services for families and children. Different teams and services that do autism assessments will help us. The investigators will ask teams and services: What speeds up diagnosis? What delays diagnosis?

The study will be in four work packages:

1. The investigators will review research in the UK and abroad to find evidence and ideas that will help speed up diagnosis.
2. The investigators will survey professionals who work for the specialist teams who diagnose autism. The survey will be about each step in the process and ask which professionals get involved. The investigators will ask about the number of children they see and the time it usually takes to reach a diagnosis. This will give us a picture of the national situation.
3. After the national survey, the investigators will select around six or eight teams. These teams will be using different and innovative approaches. The investigators will study those approaches. The investigators will talk to clinical staff, managers, referrers, parents and young people. Parents and young people will have gone through the diagnostic process. The investigators will ask parents and young people about their experiences and views. The investigators will review the steps in the diagnosis process for about 70 children in each service. The investigators will find out how long each assessment takes, how much clinical time it takes, and how much it costs. The investigators will compare findings across teams and services.
4. The investigators will have national meetings with autism experts and patient groups. The investigators will show them our findings. These groups will agree recommendations for practice. Clinical teams, service managers, commissioners, parents' groups, and NHS England will receive recommendations.

The research team has specialist expertise in autism, health services, economics, and statistics. The team includes public and NHS England partners. This will ensure the investigators take account of the needs of families and the investigators send the findings to people who plan services.

DETAILED DESCRIPTION:
Scientific Summary (following Rameses 2 reporting guidelines)

Study Title

A Realist Evaluation of Autism ServiCe Delivery (RE-ASCeD): Which diagnostic pathways work best, for whom, when, and at what cost?

Research Question Which autism diagnostic pathways work best, for whom, in what circumstances, and at what cost when providing timely and high quality diagnostic services?

Secondary Research Questions

* What factors underpin timely diagnosis service delivery success or failure?
* What needs to be in place to identify the needs and create individualized, holistic pathways of diagnosis for the child and their family?

Background The NHS England Long Term Plan states: "Children and young people with suspected autism wait too long before being provided with a diagnostic assessment. Over the next three years the investigators aim to test and implement the most effective ways to reduce waiting times…achieving timely diagnostic assessments in line with best practice guidelines...(and) to support children with autism and their families, throughout the diagnostic process." Set against a background of increasing demand for diagnostic assessment, and the need, as recommended by the NICE guidelines, for a multidisciplinary approach to assessment, taking at least 13 hours of professional time and £800 per child, evidence is needed to identify models of diagnostic assessment to achieve timely diagnoses, and how families can best be supported through this process. The NHSE Long Term Plan aims to reduce the wait time for diagnosis, and the aim of this project is to find ways/models to directly address that need.

Aims and Objectives This study aims to examine existing models of Autism diagnostic service delivery, and to investigate which approaches offer the most timely, cost-effective, high quality and child and family friendly solutions, and in line with realist thinking, to identify the factors that are likely to underpin their success, or failure, if rolled out more generally across providers.

Method

The study will use Realist Evaluation methodology, which enables evaluation of complex interventions in health care by building on existing research, to identify "what works, for whom and in what circumstances". Mixed methods, including Rapid Realist (literature) Review, survey of current practice, and case studies of centres delivering promising approaches, will be used to build a picture in an iterative manner, to identify underlying Contexts and Mechanisms that contribute to the desired Outcomes (CMO configurations) of improved Autism diagnostic service delivery and user experience, that in turn can provide plausible explanations of why the service models work or do not in certain circumstances. Data analysis from each phase of the study will be synthesised through a realist evaluative process comprising of four stages:

1. Articulation of programme theories and propositions from WP1 of the study (rapid realist review). Identification of candidate CMO configurations.
2. Data collection from WP4 (case studies) of the study to test and refine propositions.
3. Map the outcomes of each model across the cases; interrogate what contexts and mechanisms explain the pattern of outcomes.
4. Through stakeholder consolidation (WP5), refine explanatory CMO configurations to evaluate what works best and in what circumstances to deliver timely and cost-effective diagnostic services that meet the needs of children with possible Autism

Initial Programme Theory (Based on NICE principles) If there is an MDT assessment by a team with competencies in child neurodevelopment and mental health (context), then Autism will be recognised as a complex condition that relies on detailed history and observation across settings (mechanism) to diagnose it, leading to an accurate diagnosis, recognition of associated comorbidity such as ADHD and intellectual disability (outcome), and the ruling out of complex differential diagnoses.

This will also create - whilst not an explicit part of this project - accurate pictures of child strengths and needs to inform individualized packages of support and intervention through health, education and social care (outcome).

Work Package One (months 1-7). Rapid Realist Review. Evidence will be sought from published studies and evaluations of Autism diagnostic services, including controlled trials, uncontrolled studies, cost-effectiveness studies, process evaluations, grey literature and qualitative studies, including unpublished information about locally implemented Autism services. The purpose will be to refine or develop initial programme theories.

Work Package Two (months 1-6): National/International Survey of Current Diagnostic Practice: An electronic survey will be sent to UK CDCs, CAMHS teams, and tertiary centres, delivering Autism diagnostic services. This will ask teams to describe current challenges to, and any new models of diagnostic service delivery they are using. Analysis will use both qualitative and quantitative methods, to identify common themes, and services using novel approaches.

Work Package Three (months 7-9): Purposive Sampling Frame. The findings of WP 1 & 2 will be used to develop a matrix of the key features of service delivery, plus other contextual factors such as lower SES, rural, urban etc. This will be used as a sampling frame. It is anticipated that 6-8 service delivery models will be purposefully selected as case studies across the matrix to ensure the investigators have a full range of delivery models and population characteristics.

Work Package Four: Case studies (months 10-29): In-depth exploration of individual service models will be carried out to determine the interrelationship of context, intervention, mechanisms and outcomes as they occur in their natural setting. Data will be gathered within case studies using mixed methods at two levels: (i) service model and (ii) individual child/ family. Methods will include semi structured realist Interviews, focus groups, and document reviews to assemble a comprehensive description of the service and model. Interviewees will include commissioners, service managers, clinicians, referrers, parents and young people. Interviews will be recorded and transcribed, proceeding to qualitative analysis based on components of the programme theory. Regular team meetings will discuss coding, address inconsistencies, and refine collective understanding of coding framework. Coded data will be collated using NVivo software.

For each case study the journeys of at last 58 children completing the diagnostic pathway will be recorded from case notes to measure pathway, hours of professional input and time to diagnosis. Costs incurred by families for example travel to clinic, loss of earnings, will be collected by interview. Associations between service use costs and characteristics of the child and model will be assessed by regression analysis.

Work Package Five: Consolidation event, Months 27-28 : The investigators will run two iterative national consensus workshops, inviting key stakeholders including NHSE and parents/young people, to refine and confirm the context-mechanism-outcome configurations, and salient actions required to deliver timely, reliable and costed diagnostic services that meet the needs of children with possible Autism. This will lead to dissemination of models to inform the ongoing development of service models within the NHSE Long-Term Plan, commissioning guidelines and local service development.

ELIGIBILITY:
Survey Inclusion Criteria:

• Lead clinicians for childhood autism diagnostic assessment teams (children age 1-18 years), or someone who they nominate.

Survey Exclusion Criteria:

• Members of staff not involved in Autism diagnostic services.

Case Studies Inclusion Criteria :

* Parents of young people who have been through the diagnostic pathway
* Young people who have been through the diagnostic pathways
* Clinicians working in centres involved in the autism diagnostic process
* Commissioners and managers of autism services; professionals who refer in to the autism pathways

Case Studies Exclusion Criteria:

* Adults on the autism pathway
* Professionals involved in the adult autism pathway

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Members of staff. referrers, and users of Autism diagnostic services for children.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2019-11-30 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Case Study: Case Note Review - Pathway completion time taken | Up to 24 months
  Research team monitor steps in the diagnostic pathway. Access child's clinical care records for pathway completion: Time taken from referral to diagnosis/discharge (in days).

SECONDARY OUTCOMES:
Questionnaire: Reported Challenges | Up to 6 months
  National/International Survey of Current Diagnostic Practice: Asking diagnostic service teams to describe current challenges to, and any new models of diagnostic service delivery they are using.
Questionnaire: Reported Type of Service | Up to 6 months
  National/International Survey of Current Diagnostic Practice: Asking diagnostic service teams to describe type of service, e.g. Child Adolescent Mental Health Services, Child Development Clinic, Tertiary referral, in-patient ward, finance department.
Questionnaire: Reported New Models of Services | Up to 6 months
  National/International Survey of Current Diagnostic Practice: Asking diagnostic service teams to describe any new models of diagnostic service delivery they are using.
Questionnaire: Reported Geographical Area | Up to 6 months
  National/International Survey of Current Diagnostic Practice: Asking diagnostic service teams to describe Geographical area (England), e.g. population size, ethnic background, socioeconomic status.
Questionnaire: Reported Activity Levels | Up to 6 months
  National/International Survey of Current Diagnostic Practice: Asking diagnostic service teams to describe Activity levels: - Numbers of new referrals into and out of the service annually Number on current case-loads Waiting list times e.g. average Number of diagnoses (different types) per year Time taken to reach diagnosis
Questionnaire: Reported Resources Available | Up to 6 months
  National/International Survey of Current Diagnostic Practice: Asking diagnostic service teams to describe resources available:- Team size Team composition Professional multidisciplinary skill mix Facilities available Equipment available
Questionnaire: Reported Age Range of Service | Up to 6 months
  National/International Survey of Current Diagnostic Practice: Asking diagnostic service teams to describe reported age range of services
Questionnaire: Reported Clinical Remit | Up to 6 months
  National/International Survey of Current Diagnostic Practice: Asking diagnostic service teams to describe services remit and confirm type of service assessments for children for:- Autism ADHD Early trauma Neuro-disability Mental health, Common comorbidities Differential diagnoses of Autism
Questionnaire: Reported Clinical Team Competencies for Clinical Remit | Up to 6 months
  National/International Survey of Current Diagnostic Practice: Asking diagnostic service teams to describe services remit and confirm professional service competencies for children for:- Autism ADHD Early trauma Neuro-disability Mental health, Common comorbidities Differential diagnoses of Autism
Case Study - Diagnostic Team Realist Interviews | 1 hour interview during 12 month case studies
  Realist interviews either with between 6 and 12 team members per service to include commissioners, managers, clinicians, and referrers (GPs, SENCOs, HV, School nurse).
Case Study: Child and Family Interviews | 30 minutes interview during 12 month case studies
  Convenience sample of children and families who have recently been referred for assessment and diagnosis.
Case Study: Case Note Review - Dates of Meetings | Up to 20 months
  Research team monitor steps in the diagnostic pathway. Access child's clinical care records for dates of meetings to construct timeline.
Case Study: Case Note Review - Duration of Meetings | Up to 20 months
  Research team monitor steps in the diagnostic pathway. Access child's clinical care records for duration of meetings to calculate time taken overall to complete pathway.
Case Study: Case Note Review - Purpose of Clinical Meeting | Up to 20 months
  Research team monitor steps in the diagnostic pathway. Access child's clinical care records for purpose of contact with family/child for health professionals.
Case Study: Case Note Review - Test results | Up to 20 months
  Research team monitor steps in the diagnostic pathway. Access child's clinical care records for test results .
Case Study: Case Note Review Pathway completion final diagnosis | Up to 20 months
  Research team monitor steps in the diagnostic pathway. Access child's clinical care records for final diagnosis.
Case Study: Case Note Review - Pathway completion time taken | Up to 20 months
  Research team monitor steps in the diagnostic pathway. Access child's clinical care records for pathway completion: Time taken from referral to diagnosis/discharge (in days).
Case Study: Case Note Review Pathway Completion Co-Morbidities | Up to 20 months
  Research team monitor steps in the diagnostic pathway. Access child's clinical care records for any co-morbidities.
Case Study: Case Note Review Pathway Completion- type of professional involved | Up to 20 months
  Research team monitor steps in the diagnostic pathway. Access child's clinical care records for type of professionals involved.

OTHER OUTCOMES:
Realist Evaluation Outcomes | Up to 32 months
  Reported Outcomes of Autism diagnostic service delivery and user experience, that provide plausible explanations of why the service models work or do not in certain circumstances.
Realist Evaluation Contexts | Up to 32 months
  Reported Contexts of Autism diagnostic service delivery and user experience, that provide plausible explanations of why the service models work or do not in certain circumstances.
Realist Evaluation Mechanisms | Up to 32 months
  Reported Mechanisms of Autism diagnostic service delivery and user experience, that provide plausible explanations of why the service models work or do not in certain circumstances.
Rapid Realist Review | Up to 7 months
  Rapid Realist Review (RRR) will build on the systematic review undertaken in preparation of the NICE guidelines. The RRR will add to this through providing context-specific explanations for what works within a particular set of parameters. RRR is a well-established approach to synthesising evidence within a compressed time period that can identify groups of interventions or models of service delivery that relate to desired outcomes. It is also seen as consistent with the RAMESES standards for realist syntheses.
Novel Health Economic Evaluation Questionnaire: Parent Reported Experience | Every 3 months from the date of participant consent and assessed up to a maximum of 24 months
  Parents reported experience of the diagnostic process up to either diagnosis or discharge. Maximum values will be unknown until data set is complete. Reports from parents may be either positive or negative and will be on a Likert scale of 1-10 with 1 strong against the current diagnostic process and 10 strongly in favour.
Novel Health Economic Evaluation Questionnaire: Parent Reported Expenses | Every 3 months from the date of participant consent and assessed up to a maximum of 24 months
  Parents reported out of pocket expenses on travel, loss of earnings, childcare costs. Values will be in pound sterling and maximum will be unknown until data set is complete.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Male, Msc MRCP MBBCh, Principal Investigator — Sussex Community NHS Foundation Trust
Locations (1):
- Nightingale Primary Care Centre, Haywards Heath, West Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD data that is anonymised, will be released by the project steering commitee,and only then, IPD data that underlie results in publication will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting September 2023
Access Criteria: Anonymised IPD will be shared if the applicant writes to the project steering committee who will review the request. Access will only be allowed once the study is complete and all publications are complete.

REFERENCES:
- [Derived] Abrahamson V, Zhang W, Wilson PM, Farr W, Reddy V, Parr J, Peckham A, Male I. Realist evaluation of Autism ServiCe Delivery (RE-ASCeD): which diagnostic pathways work best, for whom and in what context? Findings from a rapid realist review. BMJ Open. 2021 Dec 14;11(12):e051241. doi: 10.1136/bmjopen-2021-051241. PMID 34907053
- [Derived] Abrahamson V, Zhang W, Wilson P, Farr W, Male I. Realist Evaluation of Autism ServiCe Delivery (RE-ASCeD): which diagnostic pathways work best, for whom and in what context? Protocol for a rapid realist review. BMJ Open. 2020 Jul 6;10(7):e037846. doi: 10.1136/bmjopen-2020-037846. PMID 32636288